CLINICAL TRIAL: NCT05975021
Title: A Multicenter, Randomized, Placebo-Controlled, Parallel Group Trial on the Safety and Efficacy of Istaroxime for Cardiogenic Shock SCAI Stage C
Brief Title: A Safety and Efficacy Trial of Istaroxime for Cardiogenic Shock Stage C
Acronym: SEISMiC-C
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-CL-2201; CT Id: 2023-507243-11-00 (Other: EMA)
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Istaroxime; Lactic Acid

STUDY DESIGN:
Intervention Model Description: This is a pilot, multinational, multicenter, randomized, double-blind, placebo-controlled, safety and efficacy trial. Participants will consist of males or females 18 to 85 years of age hospitalized for acute decompensated heart failure (ADHF) with persistent hypotension (systolic blood pressure [SBP] 70 to 90 mmHg for two readings with concomitant signs of hypoperfusion), and mild to moderate renal impairment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Trial treatment will be blinded to the trial staff. Istaroxime and placebo are both lyophilized powders and are put into identical vials. Each trial box will be numbered with a unique identifier, which will not allow the trial staff to ascertain which treatment is being used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Istaroxime (Experimental): Istaroxime delivered as an IV infusion via a syringe pump. Dosage regime is 1.0 µg/kg/min for 6 hours, 0.5 µg/kg/min for 42 hours. Total duration 48 hours.
  Interventions: Drug: Istaroxime
- Placebo (Placebo Comparator): Placebo (lactose) delivered as an IV infusion via a syringe pump. Total duration 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Istaroxime — IV infusion via a syringe pump. Dosage of 1.0 µg/kg/min for 6 hours; 0.5 µg/kg/min for 42 hours. Total duration 48 hours.
  Other Names: PST2744
  Arms: Istaroxime
Drug: Placebo — IV infusion via a syringe pump. Total duration 48 hours.
  Other Names: Lactate
  Arms: Placebo

SUMMARY:
The current trial aims to assess the effect of istaroxime in patients with SCAI Stage C Cardiogenic Shock (CS). These patients look unwell, frequently with a sudden change in mental status, mottled and cool extremities, and delayed capillary refill, as well as signs of congestion and relative low blood pressure and signs of hypoperfusion (reduced oxygen to organs) which frequently require support with rescue therapies including inotropes, vasopressors, or mechanical devices.

Windtree Therapeutics, Inc. has been studying istaroxime, which has the potential to treat patients in this condition without some of the disadvantages of existing therapies being used to treat patients with acute heart failure and CS.

Participants enrolled in this trial will receive standard of care (SoC) therapy for heart failure and CS. Additionally, half of the participants will be randomly chosen to receive istaroxime. Istaroxime has the potential to increase blood pressure and improve cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF);
* Clinical presentation consistent with SCAI Stage C cardiogenic shock caused by ADHF and meeting the criteria in below table;
* Admitted to ICU within 36 hours prior to randomization with congestion on chest x-ray or lung ultrasound and BNP ≥ 400 pg/mL or NT-proBNP ≥ 1400 pg/mL;
* Males and females, 18 to 85 years of age (inclusive);
* History of left ventricular ejection fraction (LVEF) ≤ 40%;
* Persistent hypotension defined as SBP between 70 and 90 mmHg for 2 readings with concomitant signs of hypoperfusion;
* Echocardiogram during initial hospitalization confirming ejection fraction ≤ 40% and no evidence of other pathology to confound interpretation of cardiac physiology (eg, pericardial effusion).

Table: Definition of SCAI Stage C Required for Inclusion. These criteria must be present at screening or prior to screening in patients actively treated by vasoactive agents or/and inotropes concomitantly (at the same time)

Must have at Least One of:

* Hypoperfusion: Venous Lactate ≥ 2 mmol/L, urine output < 30 mL/hour, cold and clammy or acute alteration in mental status.
* Hemodynamic Instability: SBP 70-90 mmHg, cardiac index < 2.2 L/min/meter2 and PCW > 15 mmHg

Without Any Of:

* Venous lactate > 5 mmol/L
* Worsening clinical status despite initial therapy (e.g., worsening hemodynamics, worsening renal or liver function)
* ALT >500 U/L (8.333 µkat/L)

Exclusion Criteria:

* Patient is in SCAI B (BP increased above 90 mmHg despite no vasoactive or inotrope therapy) or SCAI D (continuously deteriorating BP and hypoperfusion despite vasoactive or inotrope therapy);
* Lactate < 2 mmol/L (unless the patient meets the criteria in bullet 2 of Table 5-1) or lactate > 5 mmol/L prior to randomization;
* Cardiogenic shock due to any other condition besides acute decompensation of chronic heart failure;
* Any of the following in the past 30 days: acute coronary syndrome, coronary revascularization, MI, CABG, or percutaneous coronary intervention;
* Current (within 6 hours of screening) or anticipated need for treatment with renal support including ultrafiltration, or mechanical circulatory, ventilatory or renal support (intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device) such as persistent hypoperfusion and hypotension;
* History of heart transplant or UNOS priority 1a heart transplant listing
* Ongoing treatment with digoxin (if digoxin was stopped before signing the ICF and the digoxin plasma level is < 0.5 ng/ml, the patient may be enrolled);
* Severe renal impairment (eGFR < 30 ml/min, calculated by the MDRD formula);
* Hypersensitivity to the trial medication and its excipients (including known lactose hypersensitivity) or any related medication;
* Stroke or TIA within 3 months;
* Severe obstructive valvular lesions including severe aortic or mitral stenosis;
* Primary hypertrophic or restrictive cardiomyopathy or systemic illness known to be associated with infiltrative heart disease;
* Admission for AHF triggered primarily by a correctable etiology such as significant arrhythmia (inclusive of atrial fibrillation as the main reason for admission), infection, severe anemia, acute coronary syndrome, pulmonary embolism, exacerbation of COPD, planned admission for device implantation, or over-diuresis as a cause of hypotension;
* Pericardial constriction or active pericarditis;
* Significant ventricular arrhythmia prior to screening (such as sustained ventricular tachycardia or ventricular fibrillation) or implantable cardioverter defibrillator (ICD) shock within the past month or history of sudden death within 6 months;
* Cardiac resynchronization therapy (CRT), ICD, or pacemaker implantation within the past month;
* Uncontrolled arrythmia;
* Sustained hypotension (SBP < 70 mmHg) for at least 30 minutes from the time of arrival to the hospital;
* Systolic BP > 120 mmHg during the hour prior to randomization
* Cor pulmonale or other causes of isolated right-sided HF or not related to left ventricular dysfunction;
* Acute respiratory distress syndrome;
* Suspected sepsis; fever > 38° or active infection requiring IV antimicrobial treatment;
* Body weight < 40 kg or ≥ 150 kg;
* Laboratory exclusions:

  1. Hemoglobin < 9 g/dl,
  2. Platelet count < 100,000/µl,
  3. Serum potassium > 5.3 mmol/l or < 3.5 mmol/l;
* A life expectancy < 3 months based on the judgment of the investigator;
* Severe pulmonary or thyroid disease;
* Pregnant, planning on becoming pregnant, or currently breast-feeding;
* Ongoing drug or alcohol abuse;
* Participation in another interventional trial within the past 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
SBP AUC 0-6 | Start of infusion to 6 hours
  Systolic blood pressure (SBP) area under the curve (AUC) from start of infusion to 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Simonson, MD, Study Director — Windtree Therapeutics, Inc.
Locations (15):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Oregon Health and Sciences University, Portland, Oregon
- Argentina (4):
  - Sanatorio Güemes, Capital Federal, Buenos Aires
  - Sanatorio De la Trinidad Palermo, Capital Federal, Buenos Aires
  - Instituto Cardiovascular de Rosario, Rosario, Sante Fe
  - Hospital Privado de Rosario, Rosario, Sante Fe
- Kaplan Medical Center, Rehovot, Israel
- Italy (4):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - ASST degli Spedali Civili di Brescia, Brescia
  - IRCCS San Raffaele Scientific Institute, Milan
  - University of Turin, Città della Salute e della Scienza, Turin
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Uniwersytecki Szpital Kliniczny, Instytut Chorob Serca, Wroclaw
  - 4 Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
The preparation and submittal for publication of a manuscript containing the study results shall be in accordance with a process determined by a mutual written agreement between Windtree and participating institutions.
  The publication or presentation of any study results shall comply with all applicable privacy laws, including but not limited to HIPAA. This trial will be registered in the ClinicalTrials.gov and the CTIS databases, and results information from this trial will be submitted to both. In addition, every attempt will be made to publish results in peer-reviewed journals.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months after study end.
Access Criteria: Mutual written agreement.